CLINICAL TRIAL: NCT06806072
Title: EFFECTS OF BALNEOTHERAPY IN BREAST CANCER PATIENTS UNDERGOING ENDOCRINE THERAPY
Brief Title: BALNEOTHERAPY FOR BREAST CANCER PATIENTS UNDERGOING ENDOCRINE THERAPY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Parc de Salut Mar (Other)
Collaborators: Caldes de Montbui's City Council (Unknown); European Regional Development Fund (Other); Biomedical Research Networking Center on Frailty and Healthy Aging (CIBERFES) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/11531/I
Record Dates: First submitted 2025-01-23; First posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: breast cancer; balneotherapy; endocrine therapy
MeSH Terms: conditions — Breast Neoplasms | interventions — Balneology

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balneotherapy group (Experimental): These participants will be premenopausal women with estrogen receptor positive early breast cancer treated with adjuvant endocrine therapy allocated to receive 4 weeks of 3 weekly sessions of balneotherapy.
  Interventions: Other: Balneotherapy
- Control group (No Intervention): These participants will be premenopausal women with estrogen receptor positive early breast cancer treated with adjuvant endocrine therapy that will not receive balneotherapy but that will be asked to respond to the same scales and questionnaires as the balneotherapy group at the same timepoints.

INTERVENTIONS:
Other: Balneotherapy — The intervention consists in 3 weekly sessions of balneotherapy during 4 weeks.
  Arms: Balneotherapy group

SUMMARY:
Endocrine therapy is the mainstay of adjuvant therapy in premenopausal women with hormone receptive-positive (HR+) breast cancer as it has been demonstrated that it reduces long-term recurrences and increases survivial. However, this therapy, which suppresses estrogen production and estrogen-induced effects, is associated with the development of joint pain which can significantly reduce quality of life and lead to treatment discontinuation.

The main question the study aims o answer is:

Can balneotherapy (BT) alleviate muscle-skeletal pain (primary objective) derived from endocrine therapy and improve quality of life (secondary objective) in young women with HR+ breast cancer?

DETAILED DESCRIPTION:
PATIENTS AND METHODS

Inclusion Criteria:

* Premenopausal women diagnosed with early-stage hormonal receptor (HR+) breast cancer (stages I-III) undergoing ovarian suppression and aromatase inhibitor therapy (i.e., endocrine therapy) for at least three months.
* Reported musculoskeletal pain (VAS score ≥2) associated with the initiation of the endocrine therapy.

Exclusion Criteria:

* Chronic musculo-skeletal conditions predating the initiation of endocrine therapy.
* Anxiety-depression syndrome predating the initiation of endocrine therapy that is pharmacologically treated.
* Fear of water
* Fecal and urinary incontinence
* Severe venous insufficiency
* Epilepsy
* Physical disabilities that may hinder the performance of BT/aquatic exercises

Participants will be recruited in Hospital del Mar's Oncology department and in the hospital's Mineral Metabolism Clinic (Internal Medicine Department).

In addition, Caldes de Montbui's City Council will also advertise the project for patient recruitment on its public website.

Patient selection and recruitment will be performed by the study's investigators at the Hospital del Mar Research Institute.

STUDY DESIGN Prospective randomized controlled study.

STUDY FLOW Eligible particpants will undergo an initial visit (baseline) in which clinical data will be reviewed and registered. Forty-eight participants will be randomly assigned to the BT group and 48 to the control group through a lottery method. At this time point, participants will be asked to answer/complete the following scales/questionnaires: visual analog scale for pain (VAS), the SF-36 quality of life test, the Hospital Anxiety and Depression Scale (HADS), and the Pittsburgh Sleep Quality Index (PSQI). These tools measure pain severity (primary objective), quality of life, levels of anxiety and depression, and sleep quality, respectively. All results will be recorded in an anonymized database managed by the Hospital del Mar Research Institute.

Treatment Program: Participants allocated to BT group will undergo 12 sessions over four weeks (3 weekly sessions) involving thermal water exercises at 32°C (10 min inhalation, 10 min warm-up, 20 min specific exercises, 10 min relaxation), thermal showers (7 min jet or circular showers), and 30 minutes rest. Participants in the control group will be asked to not initiate new physical therapies and to continue with their usual care.

At the end of the BT program (or 4 weeks after baseline for the participants allocated to the control group), participants will be asked to answer/complete the same questionnaires/scales they did at baseline (second timepoint).

All participants will be asked to answer again the same questionnaries 6 months after BT completion or 7 months after baseline in the case of the participants of the control group (third timepoint).

Study outcomes will be obtained by calculating the differences in scores for the study variables (VAS (primary objective), SF-36, PSQI, and HADS (secondary objectives) between the end of BT and baseline, and the third timepoint vs baseline. Outcome analysis will be conducted by a qualified professional who is blinded to the two groups (BT group and control group).

In addition, the following data will be collected at baseline for each patient and included in the database for the study: age (years), Body Mass Index (BMI) (kg/m2), current medications, and time since the initiation of adjuvant endocrine therapy (months).

These data will be used as study variables and for adjustment in the multivariable analysis. The database and analyses will be managed by the principal investigator.

Data will be analyzed using descriptive statistics for qualitative variables and parametric or non-parametric tests for continuous variables. Changes in pain, quality of life, and emotional scores will be evaluated using linear models, with adjustments for confounders. Statistical significance will be set at α = 0.05.

Adverse events will be registered throughout the duration of the study. If participants allocated to the BT group report significant adverse effects directly associated with BT, they will discontinue the therapy.

ELIGIBILITY:
Inclusion Criteria:

Premenopausal women diagnosed with early-stage hormonal receptor (HR+) breast cancer (stages I-III) undergoing ovarian suppression and aromatase inhibitor therapy (i.e., endocrine therapy) for at least three months.

- Reported musculoskeletal pain (VAS score ≥2) associated with the initiation of the endocrine therapy.

Exclusion Criteria

* Chronic musculoskeletal conditions predating the initiation of endocrine therapy and/or unrelated to effects derived from the endocrine therapy (i.e. fibromyalgia)
* Anxiety-depression syndrome predating the initiation of endocrine therapy that is treated with drugs.
* Fear of water
* Fecal and/or urinary incontinence
* Severe venous insufficiency
* Epilepsy and physical disabilities that may hinder the performance of Balneotherapy (BT)/aquatic exercises.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is focused on endogen estrogenic suppression in premenopausal women so biological women are the only eligible candidates for this study.
Enrollment: 96 (Estimated)
Dates: Start 2025-02-10 (Estimated); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in musculo-skeletal pain | 7 months
  The primary objective is to determine changes in pain levels through the visual analogic scale (VAS) in the third and second timepoints vs baseline in all participants and to compare these outcomes between participants in the BT and control groups.

SECONDARY OUTCOMES:
Changes in quality of life | 7 months
  To asses changes in quality-of-life scores through the SF-36 questionnaire in the third and second timepoints vs baseline in all participants and to compare these outcomes between participants in the BT and control groups.
Changes in sleep quality | 7 months
  To asses the changes in sleep quality and sleep disturbances through the Pittsburgh Sleep Quality Index (PSQI) in the third and second timepoints vs baseline in all participants and to compare these outcomes between participants in the BT and control groups.
Changes in anxiety and depression symptoms | 7 months
  To assess the changes in anxiety and depression symptoms through the Hospital Anxiety and Depression Scale (HADS) in the third and second timepoints vs baseline in all participants and to compare these outcomes between participants in the BT and control groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Parc de Recerca Biomèdica de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No